CLINICAL TRIAL: NCT00709878
Title: Histological Characterization and Differentiation of Rash From Other EGFR Inhibitors
Brief Title: Histological Characterization and Differentiation of Rash From Other Epidermal Growth Factor Receptor (EGFR) Inhibitors
Status: Completed | Type: Observational
Sponsor: Northwestern University (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Mario Lacouture, MD, Northwestern University, Department of Dermatology
Other Study IDs: GSK-Lapatinib
Record Dates: First submitted 2008-07-01; First posted 2008-07-03 (Estimated); Results first posted 2010-09-23 (Estimated); Last update posted 2015-03-17 (Estimated); Status verified 2015-02

CONDITIONS: Skin Rash
Keywords: skin rash, lapatinib, cetuximab, erlotinib, panitumumab
MeSH Terms: conditions — Exanthema

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Skin tissue biopsies.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- L: Patients treated with lapatinib who developed skin toxicities and have been biopsied for skin rash.
  Interventions: Procedure: Skin Biopsy of Skin Rash Secondary to EGFRI Use
- C: Patients treated with cetuximab who developed skin toxicities and have been biopsied for skin rash.
  Interventions: Procedure: Skin Biopsy of Skin Rash Secondary to EGFRI Use
- P: Patients treated with panitumumab who developed skin toxicities and have been biopsied for skin rash.
  Interventions: Procedure: Skin Biopsy of Skin Rash Secondary to EGFRI Use
- E: Patients treated with erlotinib who developed skin toxicities and have been biopsied for a skin rash.
  Interventions: Procedure: Skin Biopsy of Skin Rash Secondary to EGFRI Use

INTERVENTIONS:
Procedure: Skin Biopsy of Skin Rash Secondary to EGFRI Use — Patients who were treated with lapatinib, cetuximab, panitumumab or erlotinib who subsequently developed a skin rash have been biopsied as standard of care. The biopsies will be used for this study.

SUMMARY:
The purpose of this study is to characterize the microscopic findings of skin rash associated with the use of chemotherapeutic anticancer agents known as epidermal growth factor inhibitors (EGFRIs).

DETAILED DESCRIPTION:
Epidermal growth factor (EGF) and its receptor, the EGFR, are known to be key drivers in cellular proliferation and survival. Malignant tumors result from uncontrolled cell proliferation. The use of drugs which target the EGF receptor has offered patients with non-small cell lung cancer, pancreatic cancer, head and neck cancer, and colorectal cancer additional targeted anti-cancer therapy in addition to their chemotherapeutic regimens. As a result of increased use of these EGFR inhibitors, adverse events have emerged involving the skin, hair, nails and eyes. While the EGFR inhibitors block the signal transduction that interfere with cellular proliferation and survival of cancerous cells, they also affect the normal EGF function in the skin (papulopustular rash), hair, and nails. In this study, we seek to histologically characterize the papulopustular rash in patients who have been treated with lapatinib and compare our findings with those associated with three other EGFRIs, cetuximab, erlotinib and panitumumab.

ELIGIBILITY:
Inclusion Criteria:

* Patients treated with lapatinib who developed skin toxicities and were biopsied.
* Patients treated with erlotinib, cetuximab, or panitumumab who have been biopsied for skin rash.

Exclusion Criteria:

* Patients who do not fit above criteria.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients selected for this study were treated with lapatinib, erlotinib, panitumumab or cetuximab, developed skin toxicities and were biopsied as standard of care for skin rash at the Department of Dermatology, Northwestern University.
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2008-04; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mario Lacouture, MD, Principal Investigator — Northwestern University, Department of Dermatology
Locations (1):
- Northwestern University, Chicago, Illinois, United States

REFERENCES:
- [Background] Gullick WJ. The Type 1 growth factor receptors and their ligands considered as a complex system. Endocr Relat Cancer. 2001 Jun;8(2):75-82. doi: 10.1677/erc.0.0080075. PMID 11397665
- [Background] Marmor MD, Skaria KB, Yarden Y. Signal transduction and oncogenesis by ErbB/HER receptors. Int J Radiat Oncol Biol Phys. 2004 Mar 1;58(3):903-13. doi: 10.1016/j.ijrobp.2003.06.002. PMID 14967450
- [Background] Schlessinger J. Cell signaling by receptor tyrosine kinases. Cell. 2000 Oct 13;103(2):211-25. doi: 10.1016/s0092-8674(00)00114-8. No abstract available. PMID 11057895
- [Background] Robert C, Soria JC, Spatz A, Le Cesne A, Malka D, Pautier P, Wechsler J, Lhomme C, Escudier B, Boige V, Armand JP, Le Chevalier T. Cutaneous side-effects of kinase inhibitors and blocking antibodies. Lancet Oncol. 2005 Jul;6(7):491-500. doi: 10.1016/S1470-2045(05)70243-6. PMID 15992698
- [Background] Fuchs E, Raghavan S. Getting under the skin of epidermal morphogenesis. Nat Rev Genet. 2002 Mar;3(3):199-209. doi: 10.1038/nrg758. PMID 11972157
- [Background] Lacouture ME. Mechanisms of cutaneous toxicities to EGFR inhibitors. Nat Rev Cancer. 2006 Oct;6(10):803-12. doi: 10.1038/nrc1970. PMID 16990857
- [Background] Jost M, Kari C, Rodeck U. The EGF receptor - an essential regulator of multiple epidermal functions. Eur J Dermatol. 2000 Oct-Nov;10(7):505-10. PMID 11056418
- [Background] Rodeck U, Jost M, Kari C, Shih DT, Lavker RM, Ewert DL, Jensen PJ. EGF-R dependent regulation of keratinocyte survival. J Cell Sci. 1997 Jan;110 ( Pt 2):113-21. doi: 10.1242/jcs.110.2.113. PMID 9044042
- [Background] Peus D, Hamacher L, Pittelkow MR. EGF-receptor tyrosine kinase inhibition induces keratinocyte growth arrest and terminal differentiation. J Invest Dermatol. 1997 Dec;109(6):751-6. doi: 10.1111/1523-1747.ep12340759. PMID 9406816
- [Background] Hauser PJ, Agrawal D, Hackney J, Pledger WJ. STAT3 activation accompanies keratinocyte differentiation. Cell Growth Differ. 1998 Oct;9(10):847-55. PMID 9790496
- [Background] Mimeault M, Bonenfant D, Batra SK. New advances on the functions of epidermal growth factor receptor and ceramides in skin cell differentiation, disorders and cancers. Skin Pharmacol Physiol. 2004 Jul-Aug;17(4):153-66. doi: 10.1159/000078818. PMID 15258446
- [Background] Woodworth CD, Michael E, Marker D, Allen S, Smith L, Nees M. Inhibition of the epidermal growth factor receptor increases expression of genes that stimulate inflammation, apoptosis, and cell attachment. Mol Cancer Ther. 2005 Apr;4(4):650-8. doi: 10.1158/1535-7163.MCT-04-0238. PMID 15827339
- [Background] Lorch JH, Klessner J, Park JK, Getsios S, Wu YL, Stack MS, Green KJ. Epidermal growth factor receptor inhibition promotes desmosome assembly and strengthens intercellular adhesion in squamous cell carcinoma cells. J Biol Chem. 2004 Aug 27;279(35):37191-200. doi: 10.1074/jbc.M405123200. Epub 2004 Jun 16. PMID 15205458
- [Background] Pastore S, Mascia F, Mariotti F, Dattilo C, Mariani V, Girolomoni G. ERK1/2 regulates epidermal chemokine expression and skin inflammation. J Immunol. 2005 Apr 15;174(8):5047-56. doi: 10.4049/jimmunol.174.8.5047. PMID 15814736
- [Background] Fisher GJ, Datta SC, Talwar HS, Wang ZQ, Varani J, Kang S, Voorhees JJ. Molecular basis of sun-induced premature skin ageing and retinoid antagonism. Nature. 1996 Jan 25;379(6563):335-9. doi: 10.1038/379335a0. PMID 8552187
- [Background] El-Abaseri TB, Putta S, Hansen LA. Ultraviolet irradiation induces keratinocyte proliferation and epidermal hyperplasia through the activation of the epidermal growth factor receptor. Carcinogenesis. 2006 Feb;27(2):225-31. doi: 10.1093/carcin/bgi220. Epub 2005 Aug 25. PMID 16123117
- [Background] Moy B, Goss PE. Lapatinib: current status and future directions in breast cancer. Oncologist. 2006 Nov-Dec;11(10):1047-57. doi: 10.1634/theoncologist.11-10-1047. PMID 17110623
- [Background] Albanell J, Rojo F, Averbuch S, Feyereislova A, Mascaro JM, Herbst R, LoRusso P, Rischin D, Sauleda S, Gee J, Nicholson RI, Baselga J. Pharmacodynamic studies of the epidermal growth factor receptor inhibitor ZD1839 in skin from cancer patients: histopathologic and molecular consequences of receptor inhibition. J Clin Oncol. 2002 Jan 1;20(1):110-24. doi: 10.1200/JCO.2002.20.1.110. PMID 11773160
- [Background] Busse D, Doughty RS, Ramsey TT, Russell WE, Price JO, Flanagan WM, Shawver LK, Arteaga CL. Reversible G(1) arrest induced by inhibition of the epidermal growth factor receptor tyrosine kinase requires up-regulation of p27(KIP1) independent of MAPK activity. J Biol Chem. 2000 Mar 10;275(10):6987-95. doi: 10.1074/jbc.275.10.6987. PMID 10702262
- [Background] Perez-Soler R, Delord JP, Halpern A, Kelly K, Krueger J, Sureda BM, von Pawel J, Temel J, Siena S, Soulieres D, Saltz L, Leyden J. HER1/EGFR inhibitor-associated rash: future directions for management and investigation outcomes from the HER1/EGFR inhibitor rash management forum. Oncologist. 2005 May;10(5):345-56. doi: 10.1634/theoncologist.10-5-345. PMID 15851793
- [Background] Molinari E, De Quatrebarbes J, Andre T, Aractingi S. Cetuximab-induced acne. Dermatology. 2005;211(4):330-3. doi: 10.1159/000088502. PMID 16286741
- [Background] Nelson MH, Dolder CR. Lapatinib: a novel dual tyrosine kinase inhibitor with activity in solid tumors. Ann Pharmacother. 2006 Feb;40(2):261-9. doi: 10.1345/aph.1G387. Epub 2006 Jan 17. PMID 16418322
- [Background] Cameron D. Lapatinib plus capecitabine in patients with HER2-positive advanced breast cancer. Clin Adv Hematol Oncol. 2007 Jun;5(6):456-8. No abstract available. PMID 17679920
- [Result] Nardone B, Nicholson K, Newman M, Guitart J, Gerami P, Talarico N, Yang XJ, Rademaker A, West DP, Lacouture ME. Histopathologic and immunohistochemical characterization of rash to human epidermal growth factor receptor 1 (HER1) and HER1/2 inhibitors in cancer patients. Clin Cancer Res. 2010 Sep 1;16(17):4452-60. doi: 10.1158/1078-0432.CCR-10-0421. Epub 2010 Aug 23. PMID 20732960

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 8 samples per patient/inhibitor were collected, with a total of 32 patient specimens analyzed for this study.
Groups:
- Patients Treated With Lapatinib (L): Patients treated with lapatinib who developed skin toxicities and have been biopsied for skin rash.
- Patients Treated With Cetuximab (C): Patients treated with cetuximab who developed skin toxicities and have been biopsied for skin rash.
- Patients Treated With Panitumumab (P): Patients treated with panitumumab who developed skin toxicities and have been biopsied for skin rash.
- Patients Treated With Erlotinib (E): Patients treated with erlotinib who developed skin toxicities and have been biopsied for a skin rash.
Period: Overall Study
Arm/Group | Patients Treated With Lapatinib (L) | Patients Treated With Cetuximab (C) | Patients Treated With Panitumumab (P) | Patients Treated With Erlotinib (E)
Started | 8 | 8 | 8 | 8
Completed | 8 | 8 | 8 | 8
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Patients Treated With Lapatinib (L) | Patients Treated With Cetuximab (C) | Patients Treated With Panitumumab (P) | Patients Treated With Erlotinib (E) | Total
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 32
Age, Continuous [Mean (Full Range); unit: years] | 55.7 [17 to 62] | 54.5 [34 to 72] | 65 [39 to 81] | 66.7 [46 to 81] | 60.35 [17 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 4 | 5 | 2 | 18
  Male | 1 | 4 | 3 | 6 | 14
Region of Enrollment [Number; unit: participants]
  United States | 8 | 8 | 8 | 8 | 32

OUTCOME MEASURES:

1. Primary Outcome: Differences in Histologic Alterations in Rash Caused by Lapatinib, a Dual HER1/2 Inhibitor (HER1/2i), and the Single HER1 Inhibitors (HER1i) Cetuximab, Erlotinib,and Panitumumab.
Time Frame: 6 months
Measure: Number; unit: Total number of cases
Arm/Group | Patients Treated With Lapatinib (L) | Patients Treated With Cetuximab (C) | Patients Treated With Panitumumab (P) | Patients Treated With Erlotinib (E)
Number analyzed (Participants) | 8 | 8 | 8 | 8
Total number of cases
  Ulceration | 1 | 1 | 0 | 2
  Parakeratosis | 1 | 2 | 1 | 0
  Acanthosis | 1 | 1 | 0 | 0
  Epidermal atrophy | 7 | 5 | 2 | 4
  Epidermal dysmaturation | 2 | 3 | 1 | 0
  Epidermal dyskeratosis | 3 | 3 | 0 | 0
  Epidermal neutrophilc infiltrate | 1 | 1 | 0 | 1
  Epidermal monocytic infiltrate | 0 | 0 | 2 | 0
  Epidermal eosinophilic infiltrate | 0 | 0 | 0 | 1
  Dermal neutrophilic infiltrate | 2 | 0 | 2 | 4
  Dermal monocytic infiltrate | 1 | 4 | 4 | 4
  Dermal eosinophilic infiltrate | 2 | 2 | 0 | 0
  Follicular concretions | 3 | 5 | 2 | 3
  Follicular neutrophilic pustule | 3 | 4 | 3 | 6
  Dysmorphic follicle | 4 | 2 | 2 | 4
  Follicular dyskeratosis | 4 | 3 | 1 | 1
  Follicular neurtrophilic infiltrate | 5 | 5 | 3 | 7
  Follicular monocytic infiltrate | 2 | 2 | 2 | 2
  Follicular eosinophilic infiltrate | 2 | 1 | 1 | 1
  Eccrine dyskeratosis | 0 | 1 | 0 | 0
  Eccrine necrosis | 0 | 2 | 0 | 1
  Eccrine infiltrate | 0 | 0 | 0 | 0
  Sebaceous infiltrate | 0 | 1 | 1 | 3

ADVERSE EVENTS:
Arm/Group | Patients Treated With Lapatinib (L) | Patients Treated With Cetuximab (C) | Patients Treated With Panitumumab (P) | Patients Treated With Erlotinib (E)
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 0/8 | 0/8

LIMITATIONS AND CAVEATS:
Small sample size

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No